CLINICAL TRIAL: NCT05809531
Title: An Open-Label, Nonrandomized, Multicenter Extension Study to Evaluate the Long-term Safety and Efficacy of Pegcetacoplan in Patients With C3 Glomerulopathy or Immune-Complex Membranoproliferative Glomerulonephritis
Brief Title: An Open-Label, Nonrandomized, Multicenter Extension Study to Evaluate the Long-term Safety and Efficacy of Pegcetacoplan in Participants With C3 Glomerulopathy or Immune-Complex Membranoproliferative Glomerulonephritis
Acronym: VALE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL2-C3G-314; 2023-504625-39-00 (Other: CTIS); U1111-1290-7826 (Other: Universal Trial Number (UTN)); 2022-002833-33 (EudraCT Number)
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: C3G; IC-MPGN; C3 Glomerulopathy; C3 Glomerulonephritis; Complement 3 Glomerulopathy; Complement 3 Glomerulopathy (C3G); Complement 3 Glomerulonephritis; Dense Deposit Disease; DDD; Membranoproliferative Glomerulonephritis; Membranoproliferative Glomerulonephritis (MPGN); Immune Complex Membranoproliferative Glomerulonephritis (IC-MPGN)
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative | interventions — pegcetacoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pegcetacoplan administered subcutaneously (Experimental): Pegcetacoplan administered subcutaneously twice weekly according to protocol defined dosing regimen
  Interventions: Drug: Pegcetacoplan

INTERVENTIONS:
Drug: Pegcetacoplan — Complement (C3) Inhibitor
  Other Names: APL-2

SUMMARY:
This study is designed as a long-term extension to Study APL2-C3G-310, and is being conducted to establish the long-term safety and efficacy of pegcetacoplan in patients with C3 glomerulopathy (C3G) or immune-complex membranoproliferative glomerulonephritis (IC-MPGN).

ELIGIBILITY:
Inclusion Criteria:

* Completed participation in Study APL2-C3G-310 through the week 52 visit requirements
* Experienced clinical benefit from pegcetacoplan while participating in the previous trial, in the opinion of the investigator
* Must remain on a stable regimen for C3G or IC-MPGN treatment according to the requirements of Study APL2-C3G-310
* Received vaccinations against S pneumoniae, N meningitidis (types A, C, W, Y, and B), and H influenzae (type B) according to the requirements of Study APL2-C3G-310 and agree to receive any additional vaccinations recommended according to ACIP recommendations for adults or children with complement deficiencies and/or immunocompromising conditions or other similar local applicable guidelines
* Female participants of childbearing potential, defined as any woman who has experienced menarche and who is not permanently sterile or postmenopausal, must have a negative urine pregnancy test at visit 1 and must agree to use protocol-defined methods of contraception for the duration of the study through at least 90 days after receiving the last dose of pegcetacoplan
* Male participants must agree to use protocol-defined methods of contraception and agree to refrain from donating semen for the duration of the study through at least 90 days after receiving the last dose of pegcetacoplan
* Participants above the legal age of consent, in accordance with local regulations, must be willing and able to provide informed consent. The legally authorized representative of participants under the legal age of consent must be willing and able to provide informed consent; where appropriate, participants under the legal age of consent must also give their assent to participation in the study
* Willing and able to self-administer pegcetacoplan or have an identified caregiver who can perform the administration

Exclusion Criteria:

* Female participants who are or are planning to become pregnant or who are currently breastfeeding and are unwilling to discontinue for the duration of the study and for at least 90 days after the final dose of study drug
* Inability or unwillingness to cooperate with the requirements of the protocol
* Any condition that, in the opinion of the investigator, creates an undue risk for the participant by participating in the study or is likely to confound interpretation of the study results
* Evidence of ongoing drug or alcohol abuse or dependence, in the opinion of the investigator

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with a reduction in urine protein-to-creatinine ratio (uPCR) of at least 50% from the pretreatment value over time. | 2.5 years

CONTACTS AND LOCATIONS:
Locations (47):
- United States (12):
  - Academic Medical Research Institute (01034), Los Angeles, California
  - Children's Hospital Colorado (01037), Aurora, Colorado
  - University of Florida, Department of Pediatric Nephrology (01010), Gainesville, Florida
  - Emory Investigational Drug Service (01021), Atlanta, Georgia
  - University of Iowa Hospital and Clinics (01030), Iowa City, Iowa
  - University of Michigan Hospital (01008), Ann Arbor, Michigan
  - Hackensack Meridian Health (01036), Hackensack, New Jersey
  - Cohen Children Hospital, Pediatric Pharmacy (01022), Hyde Park, New York
  - Columbia Nephrology (01039), New York, New York
  - Oregon Health & Science Univ., Dept. Pediatrics (01038), Portland, Oregon
  - Northeast Clinical Research Center LLC (01009), Bethlehem, Pennsylvania
  - Texas Children's Hospital (01027), Houston, Texas
- Argentina (2):
  - Hospital Privado-Universitario de Cordoba (54004), Córdoba
  - Clinica Privada Velez Sarsfield (54007), Córdoba
- Australia (2):
  - Kidney Trials Unit, Princess Alexandra Hospital (61007), Woolloongab, Queensland
  - St. Vincent's Hospital Melbourne (61003), Fitzroy
- Catholic University of Leuven (32001), Leuven, Belgium
- Brazil (9):
  - Santa Casa de Misericordia de Belo Horizonte (55017), Belo Horizonte, Minas Gerais
  - Irmandade da Santa Casa Misericordia Porto Alegre (55016), Porto Alegre, Rio Grande do Sul
  - HC UNESP Botucatu (55010), Botucatu
  - Hospital de Clinicas de Porto Alegre (55018), Porto Alegre
  - Real Hospital Portugues de Beneficencia (55015), Recife
  - Ruschel Medicina E Pesquisa Clinica (55012), Rio de Janeiro
  - Hospital De Base (55014), São José do Rio Preto
  - Hospital do Rim - Fundacao Oswaldo Ramos (55005), São Paulo
  - Univ Sao Paulo, Av. Dr Eneas Carvalho de Aguiar, 155 (55007), São Paulo
- Institute for Clinical and Experimental Medicine (42001), Prague, Czechia
- France (2):
  - CHU de Bordeaux - Hopital Pellegrin (33010), Bordeaux
  - Institut de transplantation urologie-nephrologie (33011), Nantes
- Schneider Childrens Medical Center (97204), Petah Tikva, Israel
- Italy (3):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico (39004), Milan
  - Istituto di Ricerche Farmacologiche Mario Negri IRCCS (39003), Ranica
  - Ospesale Pediatrico bambino Gesu (39005), Rome
- Japan (2):
  - Nagasaki University Hospital (81005), Nagasaki, Nagasaki
  - Seirei Hamamatsu General Hospital (81004), Hamamatsu, Shizuoka
- Netherlands (3):
  - AMC Apotheek Goederenontvangst (31002), Amsterdam
  - University Medical Center Groningen (31004), Groningen de Brug
  - Radboud University Medical Center (31003), Nijmegen
- South Korea (2):
  - Yonsei University College of Medicine, Sinchon Severance Hospital (82002), Seoul
  - Seoul National University Hospital (82003 & 82005), Soeul
- Spain (3):
  - Hosp. Universit. Materno-Infantil Vall d' Hebron (34006), Barcelona
  - Hospital Universitario 12 de Octubre (34008), Madrid
  - Hospital Universitario Dr Peset (34009), Valencia
- CHUV Lausanne (41002), Lausanne, Switzerland
- United Kingdom (3):
  - Imperial College Hammersmith Hospital (44013), London
  - Royal Manchester Children's Hospital (44011), Manchester
  - Nottingham University Hospitals NHS Trust (44012), Nottingham